CLINICAL TRIAL: NCT04494620
Title: Randomized Intervention Trial to Evaluate Oral Visual Inspection in the Control of Oral Cancer
Brief Title: Evaluating Oral Visual Inspection in the Control of Oral Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: Regional Cancer Centre, Trivandrum, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: RCC-IEC-Sept 2002
Record Dates: First submitted 2020-07-16; First posted 2020-07-31 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Oral Cancer
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Intervention Model Description: The control group received standard of care while the intervention group received 3 rounds of screening with visual inspection, each 3 years apart. At the 9th year of the study, once significant oral cancer mortality reduction following 3 rounds of screening among the high-risk subjects in the intervention arm was confirmed, the control arm was offered 1 round of screening with visual inspection while the intervention group was offered a 4th round of screening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (No Intervention): Standard of Care
- Intervention Arm (Active Comparator): Visual Inspection of Oral Cavity for Precancers and Cancer
  Interventions: Diagnostic Test: Visual Inspection of Oral Cavity for Precancers and Cancer

INTERVENTIONS:
Diagnostic Test: Visual Inspection of Oral Cavity for Precancers and Cancer — Participants were invited for 3 rounds of oral cavity cancer screening, conducted 3-years apart. Screening was conducted by health workers trained to perform visual inspection of the oral mucosa and identify potential precancerous lesions or oral cancer. Lesions found were referred to a weekly clinic for further evaluation by dentists and oncologists with experience in the diagnosis of oral lesions. Oral precancerous lesions were surgically excised whenever possible and those with confirmed oral cancer were referred for appropriate treatment with surgery, radiotherapy, and/or chemotherapy.
  Arms: Intervention Arm

SUMMARY:
Cluster-randomized controlled trial in Trivandrum district, Kerala, India to evaluate the effect of triennial screening for oral cavity cancer using visual inspection on oral cancer mortality.

DETAILED DESCRIPTION:
The study population consisted of 13 administrative regions (clusters) in Trivandrum district, Kerala, southern Indian. 7 clusters were randomly assigned to the intervention arm (3 rounds of oral visual inspection conducted 3 years apart) and were compared to the remaining 6 clusters assigned to a control arm that received standard of care. The eligibility criteria were all healthy subjects aged 35 and older, without a personal history of oral cancer. Informed consent was signed by each participant. The intervention arm consisted of 96,517 participants and the control group consisted of 95,356 participants.

ELIGIBILITY:
Inclusion Criteria: Residing in 13 study clusters in Trivandrum City, Kerala

Exclusion Criteria:

* Diagnosis with oral cancer prior to study
* Bedridden subjects
* Subjects suffering from open tuberculosis or other debilitating diseases

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 191873 (Actual)
Dates: Start 1996-01-01 (Actual); Primary Completion 2004-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Oral Cancer Death Rate | 15 years
  Information on all deaths were collected from the municipal and district death registers, hospital medical records, death records of churches and mosques, hospital visits by the population cancer registry staff and by project health workers. Cancer cases were coded by the ICD-O 3rd edition codes and cause of death was coded using ICD-10 by the registry and project staff blinded to study group allocation. Deaths were attributed to oral cancer if the patient had histologically or clinically confirmed oral cancer, lymph nodes or distant metastasis at the time of death or had died due to complications of oral cancer treatment.

SECONDARY OUTCOMES:
Oral Cavity Cancer Incidence | 15 years
  Information on incident oral cancer cases were obtained from the Trivandrum population-based cancer registry, hospital cancer registry of the RCC and medical records departments of other hospitals treating oral cancer patients. Collection of information was blinded to study group assignment of cases. The staging of oral cancers was done according to the UICC TNM staging system.

CONTACTS AND LOCATIONS:
Overall Officials: Kunnambath Ramadas, MD, PhD, Principal Investigator — Regional Cancer Centre, Trivandrum, India; Rengaswamy Sankaranarayanan, MD, Principal Investigator — International Agency for Research on Cancer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sankaranarayanan R, Ramadas K, Thara S, Muwonge R, Thomas G, Anju G, Mathew B. Long term effect of visual screening on oral cancer incidence and mortality in a randomized trial in Kerala, India. Oral Oncol. 2013 Apr;49(4):314-21. doi: 10.1016/j.oraloncology.2012.11.004. Epub 2012 Dec 21. PMID 23265945
- [Result] Sankaranarayanan R, Ramadas K, Thomas G, Muwonge R, Thara S, Mathew B, Rajan B; Trivandrum Oral Cancer Screening Study Group. Effect of screening on oral cancer mortality in Kerala, India: a cluster-randomised controlled trial. Lancet. 2005 Jun 4-10;365(9475):1927-33. doi: 10.1016/S0140-6736(05)66658-5. PMID 15936419
- [Derived] Cheung LC, Ramadas K, Muwonge R, Katki HA, Thomas G, Graubard BI, Basu P, Sankaranarayanan R, Somanathan T, Chaturvedi AK. Risk-Based Selection of Individuals for Oral Cancer Screening. J Clin Oncol. 2021 Feb 20;39(6):663-674. doi: 10.1200/JCO.20.02855. Epub 2021 Jan 15. PMID 33449824